CLINICAL TRIAL: NCT03659578
Title: A Phase II Study of Thymopeptide a1 During Split-course Chemoradiotherapy to Reduce Acute Pneumonia For Bulky None-small Cell Lung Cancer
Brief Title: Study of Thymosin α1 to Reduce Acute Pneumonia For Bulky None-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1043
Record Dates: First submitted 2018-09-02; First posted 2018-09-06 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Split-course Chemoradiotherapy; Thymosin a1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thymalfasin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thymosin α1 (Experimental): Patients are treated with subcutaneous injections of thymosin once a week,1.6mg each time from the start of radiation to 2 months after the end of radiation.
  Interventions: Drug: Concurrent chemotherapy; Radiation: split-course radiotherapy; Drug: thymosin alpha 1

INTERVENTIONS:
Drug: Concurrent chemotherapy — Concurrent chemotherapy consists of weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡), each of 1 day's duration.
Radiation: split-course radiotherapy — Patient was administered with 51 Gy in 17 fractions or 40 Gy in 10 fractions as the first course followed by a break of four weeks. Patients without disease progression had a dose of 15 Gy in 5 fractions or 24 Gy in 6 fractions as a boost
Drug: thymosin alpha 1 — subcutaneous injections of thymosin once a week,1.6mg each time from the start of radiation to 2 months after the end of radiation.

SUMMARY:
This Phase II study is to determine the efficacy of Thymosin α1 on the frequency of acute pneumonia in non-small cell lung cancer with bulky tumor.

DETAILED DESCRIPTION:
This Phase II study is to determine the efficacy of Thymosin α1 on the frequency of radiation pneumonitis in non-small cell lung cancer with bulky tumor.

All patients received four cycles of weekly docetaxel (25mg/㎡) and nedaplatin (25mg/㎡)(DP), each of 1 day's duration, combined with split-course thoracic radiotherapy of 51 Gy in 17 fractions or 40 Gy in 10 fractions as the first course followed by a break of four weeks. Patients without disease progression had a dose of 15 Gy in 5 fractions or 24 Gy in 6 fractions as a boost. Patients were further treated with subcutaneous injections of thymosin once a week,1.6mg each time from the start of radiation to 2 months after the end of radiation. Toxicities will be graded according to CTCAE v. 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of NSCLC.
* Patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

  * Unresectable phase IIIA-IIIC lung cancer confirmed by PET/CT, CT or MRI.
  * Whole lung V20>=35% when giving 60Gy which is the minimum dose of radical irradiation.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Previously treated with chemotherapy or treatment-naive
* No previous chest radiotherapy, immunotherapy or biotherapy
* Hemoglobin≥10 mg/dL, platelet≥100000/μL,absolute neutrophil count ≥1500/μL
* Serum creatinine ≤1.25 times the upper normal limit(UNL), or creatinine clearance≥60 ml/min
* Bilirubin ≤1.5 times UNL, AST（SGOT）≤2.5 times UNL ,ALT（SGPT）≤2.5 times UNL,alkaline phosphatase ≤5 times UNL
* FEV1 >0.8 L
* CB6 within normal limits
* patients and their family signed the informed consents

Exclusion Criteria:

* Previous or recent another malignancy, except nonmelanoma skin cancer or cervical cancer in situ
* Contraindication for chemotherapy
* Malignant pleural or pericardial effusion.
* Women in pregnancy, lactation period, or no pregnancy test 14 days before the first dose
* Women who has the probability of pregnancy without contraception
* Tendency of hemorrhage
* In other clinical trials within 30 days
* Addicted in drugs or alcohol, AIDS patients
* Uncontrollable seizure or psychotic patients without self-control ability
* Severe allergy or idiosyncrasy
* Not suitable for this study judged by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of ≥grade 2 radiation pneumonitis (CTCAE 5.0 version) | 1-year
  Radiation-induced pneumonitis except other reasons induced pneumonia

SECONDARY OUTCOMES:
Total lymphocyte count | From the beginning of CCRT until 6 months after the completion of CCRT.
C-reaction protein | From the beginning of CCRT until 6 months after the completion of CCRT.
grade of pulmonary fibrosis (CTCAE 5.0 version) | 1-year

OTHER OUTCOMES:
Alpha diversity of gut microbiota as the exploratory outcome | From baseline to the end of CCRT, an average of 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Mery B, Guy JB, Swalduz A, Vallard A, Guibert C, Almokhles H, Ben Mrad M, Rivoirard R, Falk AT, Fournel P, Magne N. The evolving locally-advanced non-small cell lung cancer landscape: Building on past evidence and experience. Crit Rev Oncol Hematol. 2015 Nov;96(2):319-27. doi: 10.1016/j.critrevonc.2015.05.020. Epub 2015 Jun 7. PMID 26095618
- [Background] Furuse K, Fukuoka M, Kawahara M, Nishikawa H, Takada Y, Kudoh S, Katagami N, Ariyoshi Y. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with mitomycin, vindesine, and cisplatin in unresectable stage III non-small-cell lung cancer. J Clin Oncol. 1999 Sep;17(9):2692-9. doi: 10.1200/JCO.1999.17.9.2692. PMID 10561343
- [Background] Wang T, Nelson RA, Bogardus A, Grannis FW Jr. Five-year lung cancer survival: which advanced stage nonsmall cell lung cancer patients attain long-term survival? Cancer. 2010 Mar 15;116(6):1518-25. doi: 10.1002/cncr.24871. PMID 20108308
- [Background] Curran WJ Jr, Paulus R, Langer CJ, Komaki R, Lee JS, Hauser S, Movsas B, Wasserman T, Rosenthal SA, Gore E, Machtay M, Sause W, Cox JD. Sequential vs. concurrent chemoradiation for stage III non-small cell lung cancer: randomized phase III trial RTOG 9410. J Natl Cancer Inst. 2011 Oct 5;103(19):1452-60. doi: 10.1093/jnci/djr325. Epub 2011 Sep 8. PMID 21903745
- [Background] Fournel P, Robinet G, Thomas P, Souquet PJ, Lena H, Vergnenegre A, Delhoume JY, Le Treut J, Silvani JA, Dansin E, Bozonnat MC, Daures JP, Mornex F, Perol M; Groupe Lyon-Saint-Etienne d'Oncologie Thoracique-Groupe Francais de Pneumo-Cancerologie. Randomized phase III trial of sequential chemoradiotherapy compared with concurrent chemoradiotherapy in locally advanced non-small-cell lung cancer: Groupe Lyon-Saint-Etienne d'Oncologie Thoracique-Groupe Francais de Pneumo-Cancerologie NPC 95-01 Study. J Clin Oncol. 2005 Sep 1;23(25):5910-7. doi: 10.1200/JCO.2005.03.070. Epub 2005 Aug 8. PMID 16087956
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Marks LB, Bentzen SM, Deasy JO, Kong FM, Bradley JD, Vogelius IS, El Naqa I, Hubbs JL, Lebesque JV, Timmerman RD, Martel MK, Jackson A. Radiation dose-volume effects in the lung. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S70-6. doi: 10.1016/j.ijrobp.2009.06.091. PMID 20171521
- [Background] Gielda BT, Marsh JC, Zusag TW, Faber LP, Liptay M, Basu S, Warren WH, Fidler MJ, Batus M, Abrams RA, Bonomi P. Split-course chemoradiotherapy for locally advanced non-small cell lung cancer: a single-institution experience of 144 patients. J Thorac Oncol. 2011 Jun;6(6):1079-86. doi: 10.1097/JTO.0b013e3182199a7c. PMID 21532501
- [Background] Spoelstra FO, Pantarotto JR, van Sornsen de Koste JR, Slotman BJ, Senan S. Role of adaptive radiotherapy during concomitant chemoradiotherapy for lung cancer: analysis of data from a prospective clinical trial. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1092-7. doi: 10.1016/j.ijrobp.2008.12.027. Epub 2009 Mar 26. PMID 19327915
- [Background] Dang J, Li G, Ma L, Diao R, Zang S, Han C, Zhang S, Yao L. Predictors of grade >/= 2 and grade >/= 3 radiation pneumonitis in patients with locally advanced non-small cell lung cancer treated with three-dimensional conformal radiotherapy. Acta Oncol. 2013 Aug;52(6):1175-80. doi: 10.3109/0284186X.2012.747696. Epub 2012 Dec 3. PMID 23198719
- [Background] Ji K, Zhao LJ, Liu WS, Liu ZY, Yuan ZY, Pang QS, Wang J, Wang P. Simultaneous integrated boost intensity-modulated radiotherapy for treatment of locally advanced non-small-cell lung cancer: a retrospective clinical study. Br J Radiol. 2014 Mar;87(1035):20130562. doi: 10.1259/bjr.20130562. Epub 2014 Jan 27. PMID 24588668
- [Background] McDonald S, Rubin P, Phillips TL, Marks LB. Injury to the lung from cancer therapy: clinical syndromes, measurable endpoints, and potential scoring systems. Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1187-203. doi: 10.1016/0360-3016(94)00429-O. PMID 7713782
- [Background] Barthelemy-Brichant N, Bosquee L, Cataldo D, Corhay JL, Gustin M, Seidel L, Thiry A, Ghaye B, Nizet M, Albert A, Deneufbourg JM, Bartsch P, Nusgens B. Increased IL-6 and TGF-beta1 concentrations in bronchoalveolar lavage fluid associated with thoracic radiotherapy. Int J Radiat Oncol Biol Phys. 2004 Mar 1;58(3):758-67. doi: 10.1016/S0360-3016(03)01614-6. PMID 14967431
- [Background] Trott KR, Herrmann T, Kasper M. Target cells in radiation pneumopathy. Int J Radiat Oncol Biol Phys. 2004 Feb 1;58(2):463-9. doi: 10.1016/j.ijrobp.2003.09.045. PMID 14751516
- [Background] Rasmussen L, Arvin A. Chemotherapy-induced immunosuppression. Environ Health Perspect. 1982 Feb;43:21-5. doi: 10.1289/ehp.824321. PMID 7037385
- [Background] Brambilla C, Romand P, Vanderkerckhove C, Moro D. [Respiratory infection and bronchial cancer]. Rev Mal Respir. 1992;9 Suppl 1:R49-52. French. PMID 1317051
- [Background] Klastersky J. [The infectious complications of bronchial cancer]. Rev Mal Respir. 1998 Sep;15(4):451-9. French. PMID 9805755
- [Background] Zhuang H, Yuan Z, Chang JY, Wang J, Pang Q, Zhao L, Wang P. Radiation pneumonitis in patients with non--small-cell lung cancer treated with erlotinib concurrent with thoracic radiotherapy. J Thorac Oncol. 2014 Jun;9(6):882-5. doi: 10.1097/JTO.0000000000000126. PMID 24828665
- [Background] Wu J, Zhou L, Liu J, Ma G, Kou Q, He Z, Chen J, Ou-Yang B, Chen M, Li Y, Wu X, Gu B, Chen L, Zou Z, Qiang X, Chen Y, Lin A, Zhang G, Guan X. The efficacy of thymosin alpha 1 for severe sepsis (ETASS): a multicenter, single-blind, randomized and controlled trial. Crit Care. 2013 Jan 17;17(1):R8. doi: 10.1186/cc11932. PMID 23327199
- [Background] Romani L, Bistoni F, Gaziano R, Bozza S, Montagnoli C, Perruccio K, Pitzurra L, Bellocchio S, Velardi A, Rasi G, Di Francesco P, Garaci E. Thymosin alpha 1 activates dendritic cells for antifungal Th1 resistance through toll-like receptor signaling. Blood. 2004 Jun 1;103(11):4232-9. doi: 10.1182/blood-2003-11-4036. Epub 2004 Feb 24. PMID 14982877
- [Background] Zheng BX, Cheng DY, Xu G, Fan LL, Yang Y, Yang W. [The prophylactic effect of thymosin alpha 1 on the acute exacerbation of chronic obstructive pulmonary disease]. Sichuan Da Xue Xue Bao Yi Xue Ban. 2008 Jul;39(4):588-90. Chinese. PMID 18798500
- [Background] Zatloukal P, Petruzelka L, Zemanova M, Havel L, Janku F, Judas L, Kubik A, Krepela E, Fiala P, Pecen L. Concurrent versus sequential chemoradiotherapy with cisplatin and vinorelbine in locally advanced non-small cell lung cancer: a randomized study. Lung Cancer. 2004 Oct;46(1):87-98. doi: 10.1016/j.lungcan.2004.03.004. PMID 15364136
- See also: 11. National Comprehensive Cancer Network. (NCCN) Clinical Practice Guidelines in Oncology. Small Cell Lung Cancer, Version — https://www.nccn.org/professionals/physician_gls/f_guidelines.asp